CLINICAL TRIAL: NCT04627636
Title: Myofascial Trigger Points Release With Shockwave Therapy on Pain and Function of Shoulder Hand Syndrome in Stroke Patients With Diabetic Neuropathy
Brief Title: MTPr With Shockwave on Pain & Function of SHS in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Lama Saad El-Din Mahmoud, Lecturer of physical therapy, Department of Neuromuscular disorders and its surgery, faculty of physical therapy, october 6 univerisity, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No: P.T.REC/012/002459
Record Dates: First submitted 2020-11-08; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Stroke
Keywords: Stroke; Diabetic Neuropathy; Shoulder hand syndrome
MeSH Terms: conditions — Stroke; Diabetic Neuropathies; Reflex Sympathetic Dystrophy | interventions — Drainage

STUDY DESIGN:
Intervention Model Description: study group: which treated with MTrPs release combined with shockwave therapy and conventional program, while control group: treated with a conventional selected exercise program
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): which treated with MTrPs release combined with shockwave therapy and conventional program
  Interventions: Other: Myofascial trigger points pressure (MTrP) release; Other: Shockwave therapy application; Other: conventional therapy
- control group (Experimental): which treated with conventional physical therapy program
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: Myofascial trigger points pressure (MTrP) release — Myofascial trigger points pressure (MTrP) release technique, the initial step was to recognize and find the trigger points (TP) , and The second step after TP palpation was the MTrP release technique, as follow, by one or both hands, the thumbs or four fingers of the therapist applied a maintained pressure, pushing internal toward the middle
  Arms: study group
Other: Shockwave therapy application — The JEST-2000 (JOEUN Medical, Dae-Jeon, South Korea) was used for the ESWT. The application of pressure pulses of ESWT was centered around the flexor muscles with hypertonia
  Arms: study group
Other: conventional therapy — Passive ROM exercises performed by the therapist and Bobath Neurodevelopmental Approach (prolonged stretch): The Intervention methods for Bobath involved the activation of key points of control for the reduction of tone

SUMMARY:
Background: shoulder-hand syndrome is considered a significant reason for the reduction of upper limb functions after stroke. Purpose: To investigate the influence of Myofascial Trigger Points (MTrPs) release and shockwave therapy on pain and functions of the upper extremity in stroke patients with diabetic neuropathy.

DETAILED DESCRIPTION:
Methods: two equal groups of thirty stroke patients, divided into, study group: which treated with MTrPs release combined with shockwave therapy and conventional program, while control group: treated with a conventional selected exercise program.

ELIGIBILITY:
Inclusion Criteria:

* stroke from 4:8 months
* age ranging from 45:60 years
* All the patients were identified with SHS as diagnosed by the Diagnostic criteria for SHS post-stroke 18 and were in stage I of syndrome evolution

Exclusion Criteria:

* any other causes of shoulder pain in the hemiplegic side of the body
* a cognitive impairment
* structured joint deformity in the painful shoulder or hand
* other musculoskeletal disorders of UE.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
- Complex Regional Pain Syndrome (CRPS) severity score | 4 weeks
  It is a quantitative index and valid instrument to score and monitor the severity of CRPS and SHS.
- Figure-of-Eight Method of Measuring Hand Size for hand swelling | 4 weeks
  The figure-of-eight technique utilizing tape measurement for hand size
- Visual analogue scale for pain (VAS-P) for pain assessment | 4 weeks
  The VAS for pain is a valid and reliable assessment of pain intensity, as a straight horizontal line of fixed length (10 cm) considered the simplest VAS.

CONTACTS AND LOCATIONS:
Locations (1):
- Lama S Mahmoud, Al Jīzah, Select State, Egypt